CLINICAL TRIAL: NCT00161109
Title: Genetics and Psychopathology in the 22q11 Deletion Syndrome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: UMC Utrecht (Other)
Collaborators: Netherlands Brain Foundation (Other); Children's Hospital of Philadelphia (Other)
Other Study IDs: P03.0377C
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2006-10-13 (Estimated); Status verified 2004-10

CONDITIONS: Chromosome 22q11.2 Deletion Syndrome
Keywords: 22q11.2 deletion syndrome; Psychopathology; Psychiatry; Neuropsychology; Psychiophysiology; Autism; Psychosis; Deletion size; Candidate genes; Psychiatric symptoms; Neuropsychological impairments; Psychophysiological performance
MeSH Terms: conditions — DiGeorge Syndrome; Autistic Disorder; Psychotic Disorders

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
The purposes of this study are to:

1. study the nature and longitudinal course of psychiatric symptoms in children with the 22q11.2 deletion syndrome and
2. identify genes that contribute to the occurrence of these symptoms.

DETAILED DESCRIPTION:
The study of genes that are implicated in various mental diseases is increasingly relevant. The association between a gene and a disease can provide valuable information on how the neurobiology of the brain is altered, by studying the function of the protein encoded by the gene. This information is important for the development of new treatments.

However, the identification of these "disease" genes is difficult, due to the complexity of human behavior and the interaction of multiple genes. Moreover, the human genome consists of approximately 35,000 genes, further complicating the matter.

The situation is simplified when a psychiatric disorder and a genetic anomaly co-occur; assuming a causative relation, one can focus on the implicated genetic region.

The 22q11-deletion syndrome (22q11DS) is an example of this type; this syndrome is caused by a disappearance ("deletion") of 20-30 genes in a well-defined region on chromosome 22. People with 22q11DS have a high risk of autism and psychosis, therefore one or more genes in the 22q11DS region must be associated with these disorders.

In this study we aim to identify these genes, by carefully studying psychiatric symptoms (and additional parameters of brain functioning) in a large sample of 22q11DS children and subsequently statistically correlate these findings to specific genes within the 22q11DS region. If genes associated with autism and/or psychosis in the 22q11DS population can be found, they may help to understand the underlying neurobiology that cause these diseases, not only in 22q11DS patients but in the general population as well.

The aims of this study are:

1. STUDY NATURE AND DEVELOPMENTAL COURSE OF PSYCHIATRIC SYMPTOMS. To perform a prospective longitudinal follow up study of a sample of children with the 22q11.2 deletion syndrome with specific attention to a) possible predictors for psychosis in psychiatric and neuropsychological profile and b) a possible correlation between autistic symptoms and psychosis.
2. ASSESS THE CORRELATION OF 22q11.2 DELETIONS WITH THE PSYCHOSIS / AUTISTIC PHENOTYPE AND ASSOCIATED ENDOPHENOTYPES: To evaluate whether the size of the deletion and / or polymorphisms at selected candidate genes within the 22q11.2 deleted region contribute to the psychosis and or autistic phenotype or to related psychophysiologic / neuropsychological impairments in 22q11DS.

METHODS.

With regard to aim 1:

A large sample (a final sample size of 100-120 is anticipated) of children with 22q11DS, aged 10 - 20 year, is broadly phenotyped using standard psychiatric assessment methods, intelligence and selected neuropsychological tests as well as psychophysiological assessments. Approximately 4 years after the initial assessment a follow up assessment is planned. Age and IQ matched children without the deletion (or any other apparent genetic abnormality) are used as a control group.

With regard to aim 2:

* Phenotypes: Individuals with a certain endophenotype ("cases" e.g. the presence of autistic symptoms or a decreased Pre Pulse Inhibition or impaired performance on executive tasks) will be compared to children without that particular phenotype ("controls").
* Genetic analysis:

  * Genotyping consists of:

    1. assessment of the size of the deletion and
    2. genotyping single nucleotide polymorphisms (SNPs) across the deleted genomic region. Genotyping will be performed using approximately 75 previously characterized SNPs, with an increased density of SNPs in the target candidate genes (~3-5 SNPs per candidate gene). In order to determine whether a haplotype and/or variants of genes within region 22q11.2 contribute to the autistic phenotype and related neuro-psychological impairments in patients with the deletion, we will identify DNA polymorphisms using existing databases. We will then genotype patients with the 22q11.2 deletion for the selected polymorphisms and compare the allele frequencies and haplotype combinations in 22q11DS patients with the phenotype ("cases") to those deleted patients without these findings ("controls") applying chi-square, Fisher's exact test, and other statistical genetic methods as appropriate.

ELIGIBILITY:
Inclusion Criteria:

* 22q11.2 deletion confirmed with fluorescence in-situ hybridization (FISH)

Exclusion Criteria:

* None

Ages: 8 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 175
Dates: Start 2002-10; Study Completion 2012-10

CONTACTS AND LOCATIONS:
Overall Officials: René S. Kahn, M.D., Ph.D., Study Director — UMC Utrecht, The Netherlands
Locations (2):
- Children's Hospital of Philadelphia, Dpt of Genetics and Dpt of Child and Adolescent Psychiatry, Philadelphia, Pennsylvania, United States
- UMC Utrecht, Dpt of Child and Adolescent Psychiatry, Utrecht, Netherlands